CLINICAL TRIAL: NCT07059039
Title: Impact of Antibio Prophylaxis on Occurence of Ventilator Associated Pneumonia in Trauma Patients
Acronym: antiVAP
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240894
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-07

CONDITIONS: Ventilator Associated Pneumonia ( VAP)
Keywords: trauma; antibioprophylaxis; pneumonia; ventilator associated pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated; Wounds and Injuries; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Early antibiotic prophylaxis group: Group will consist of patients meeting the inclusion criteria and :
  * in whom systemic intravenous antibiotic prophylaxis has been initiated within 24 hours of the start of medical management
  * with a duration of systemic antibiotic prophylaxis of between 24h and 72h
- Control group: The group will be made up of patients meeting the inclusion criteria and :
  - in whom no systemic antibiotic prophylaxis (apart from any intraoperative antibiotic prophylaxis) was administered during the first 72 hours after the start of medical care

SUMMARY:
The relevance of a short course of antibiotic prophylaxis for the prevention of ventilator assocaited pneumonia (VAP) in trauma patients, and its impact on bacterial ecology, remains to be clarified.

Antibiotics are often administered in the pre-hospital phase, usually in cases to traumatic lesions with high risk of secondary infection (open fractures, deteriorating wounds, etc.). If there is a potential benefit of such antibiotic prophylaxis on the risk of surgical site infection, there could also be a benefit on the risk of developing pulmonary infections. Recent data have shown a reduction in the risk of early-onset VAP in cerebrovascular patients with a strategy of very early administration of antibiotic prophylaxis (PROPHYVAP study(1)), as well as in patients taken into intensive care following cardiac arrest (ANTHARTIC study(2)). The aim of the study is to evaluate the impact of early systemic antibiotic prophylaxis in trauma patients on the incidence of early VAP during the ICU stay.

DETAILED DESCRIPTION:
VAP is the most frequent infectious complication in the Intensive Care Units (ICU), with a higher incidence in trauma patients.

Individually, the development of VAP prolongs the duration of mechanical ventilation and in-hospital lenghts of stay, and is associated with additional costs. Collectively, VAP is responsible for around half of all antibiotic consumption in the ICU, with ecological consequences through the emergence of bacterial resistance. Numerous studies and recommendations have been published on the prevention of VAPs. According to current recommendations, this prevention is based on a standardized multimodal approach, including systematic digestive decontamination (SDD) combining an enteral topical antiseptic and systemic antibiotic prophylaxis for less than 5 days to reduce mortality. However, the application of SDD remains limited, and few recent studies have focused on trauma patients. Recently, several studies and meta analysis showed a patential benefit of a single short course of systemic antibiotics (not full SDD) on the risk of subsequent VAP, especially in brain injured patients. The value of short-term antibiotic prophylaxis in trauma patients therefore remains to be documented. The aim of this study is to evaluate the impact of early antibiotic prophylaxis on the risk of VAP in a population of severe trauma patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Trauma patient: admitted between 01/01/2021 and 31/12/2023 for suspected severe trauma (included in TraumaBase® )
* Put on mechanical ventilation during the first 24 hours following the start of medical care (including pre-hospital care)
* Patient on MV for at least 48 consecutive hours during intensive care stay
* Patient does not object to the use of his/her data for this research

Exclusion Criteria:

* Patient under full selective digestive decontamination protocol
* Early inhaled antibiotic prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult trauma patients placed on mechanical ventilation during the first 24 hours of management, and for a duration of at least 48 hours
Sampling Method: Non-Probability Sample
Enrollment: 2143 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
early onset ventilator associated pneumonia (VAP) | 28 days after ICU admission
  Incidence of early onset VAP (≤ 7 days after mechanical ventilation)

SECONDARY OUTCOMES:
incidence of VAP | 28 days after ICU admission
  Incidence of VAP, whatever the dely of occurrence
Incidence of late onset VAP | 28 days after ICU admission
  Incidence of late onset VAP (>7 days after mecahnical ventilation)
number of VAP | 28 days after ICU admission
  number of VAP during ICU stay
Incidence of non-respiratory sepsis | 28 days after ICU admission
  Incidence of non-respiratory sepsis during ICU stay
Incidence of surgical site infection | 28 days after ICU admission
  Incidence of surgical site infection during ICU stay
acquisition of multidrug resistant bacteria | 28 days after ICU admission
  acquisition of MDR bacteria during ICU stay
number of days with mechanical ventilation | 28 days after ICU admission
  Number of days with mechanical ventilation during ICU stay
length of ICU stay | 28 days after ICU admission
  length of ICU stay
length of hospital stay | 28 days after ICU admission
  length of hospital stay
mortality at 28 days | 28 days after ICU admission
  mortality at 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Arnaud Foucrier, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Beaujon, Clichy, France

REFERENCES:
- [Background] Dahms K, Ansems K, Dormann J, Steinfeld E, Janka H, Metzendorf MI, Breuer T, Benstoem C. Effectiveness of antibiotic prophylaxis in polytrauma patients: a systematic review and meta-analysis. Eur J Trauma Emerg Surg. 2025 Feb 13;51(1):105. doi: 10.1007/s00068-025-02789-8. PMID 39945862
- [Background] Hadley-Brown K, Hailstone L, Devane R, Chan T, Devaux A, Davis JS, Hammond N, Li Q, Litton E, Myburgh J, Poole A, Santos J, Seppelt I, Tong SYC, Udy A, Venkatesh B, Young PJ, Delaney AP. Prophylactic Antibiotics in Adults With Acute Brain Injury Who Are Invasively Ventilated in the ICU: A Systematic Review and Meta-Analysis. Chest. 2025 Apr;167(4):1079-1089. doi: 10.1016/j.chest.2024.10.031. Epub 2024 Oct 28. PMID 39490972
- [Background] Dahyot-Fizelier C, Lasocki S, Kerforne T, Perrigault PF, Geeraerts T, Asehnoune K, Cinotti R, Launey Y, Cottenceau V, Laffon M, Gaillard T, Boisson M, Aleyrat C, Frasca D, Mimoz O; PROPHY-VAP Study Group and the ATLANREA Study Group. Ceftriaxone to prevent early ventilator-associated pneumonia in patients with acute brain injury: a multicentre, randomised, double-blind, placebo-controlled, assessor-masked superiority trial. Lancet Respir Med. 2024 May;12(5):375-385. doi: 10.1016/S2213-2600(23)00471-X. Epub 2024 Jan 20. PMID 38262428